CLINICAL TRIAL: NCT04550663
Title: One-center, Open-label, Single-arm Clinical Study of the Safety and Effectiveness of NKG2D CAR-T Cells Infusion in the Treatment of Relapsed/ Refractory NKG2DL+ Tumors
Brief Title: NKG2D CAR-T(KD-025) in the Treatment of Relapsed or Refractory NKG2DL+ Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: KAEDI (Other)
Responsible Party: Principal Investigator, Baorui Liu, Professor of Medicine, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-172-01
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumor; Hepatocellular Carcinoma; Colorectal Cancer; Glioma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD-025 CAR-T cells (Experimental): NKG2D-based CAR-T cells infusion
  Interventions: Drug: KD-025 CAR-T cells

INTERVENTIONS:
Drug: KD-025 CAR-T cells — Autologous genetically modified anti-NKG2DLs CAR transduced T cells

SUMMARY:
This is a Phase 1, single-arm, single-center, open-label study to evaluate the safety and effectiveness of NKG2D-based CAR-T cells infusion in the treatment of relapsed/refractory NKG2DL+ solid tumors.

DETAILED DESCRIPTION:
In this study,the enrollment of the patients must meet the inclusion and exclusion criteria . All subjects will be asked to continue to undergo long-term gene safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, male & female;
2. Patients with recurrent/refractory NKG2DL+ tumors diagnosis by pathological histology or cytology, focus on the inclusion of patients with hepatocellular carcinoma positive. (If recruit liver cancer patients, patients should with locally advanced or metastatic hepatocellular carcinoma (HCC), Barcelona clinic liver cancer (BCLC) staging system classification for B or C, for B, patients are not suitable for local treatment and/or surgery, or disease progression occurs after surgery and/or local treatment, or declined to surgery and/or local treatment);
3. Patients who fail first-line treatment or are unwilling to receive first-line treatment;
4. Disease progression occurred within 14 days before inclusion (RECIST criteria must be used as a basis for assessment of disease progression). According to RECIST V1.1, patients have at least one measurable lesion. Target lesions located within the field of previous therapeutic irradiation or within the area of local treatment (interventional or ablative treatment) are considered measurable if progress is confirmed;
5. The main organs function normally and meet the following requirements;

   Blood routine examination shall be in accordance with (no blood transfusion within 14 days) :
   1. HB≥90g/L
   2. ANC ≥1.5×10^9/L
   3. PLT ≥75×10^9/L

   serum biochemicals examination shall be in accordance with:
   1. BIL <1.5 upper normal limit (ULN)
   2. ALT and AST<2.5×ULN; In the case of liver metastasis, ALT and AST<5×ULN
   3. Serum Cr≤1×ULN, endogenous creatinine clearance≥50ml/min(Cockcroft-Gault formula)；
6. ECOG physical condition score: 0-1;
7. Expected survival time ≥3 months;
8. Cardiac function well before inclusion, no myocardial infarction attack occurred within half a year, and hypertension and other coronary heart disease were under control at present;
9. No other uncontrollable benign diseases such as lung, kidney, liver infection before enrollment;
10. Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 7 days of enrollment and voluntarily use an appropriate method of contraception during observation and within 8 weeks after the last administration; men should be surgically sterilized or agree to use an appropriate method of contraception during the observation period and within 8 weeks after the last administration;
11. Patients voluntarily participated in this trial and sign the informed consent form;
12. Patients with compliance and expected to follow up the efficacy and adverse reactions as required by the protocol；
13. CAR-T cells amplify successfully to the expected number.

Exclusion Criteria:

1. Pregnant or lactating women, pregnancy test positive by blood or urine within 48 hours before immune cell transplantation;
2. Patients who need to be treated with systemic steroid;
3. Under following treatment conditions currently:

   1. during the other anti-tumor clinical observation period within 14 days before blood collection;
   2. patient has not recovered from acute side effects of the previous treatment;
4. Receive radiotherapy within 4 weeks before enrollment;
5. Patients who received any other cell therapy before;
6. Transfection efficiency of lymphocytes of patients < 5% in feasibility assessment screening stage, or T cell amplification efficiency < 5 times；
7. Uncontrolled symptoms or other illnesses, including but not limited to infection, congestive heart failure, unstable angina, arrhythmia, psychosis;
8. Patients with severe acute allergic reactions, or the attending doctor believes there is an unpredictable risk;
9. Patients who have received other cell therapies;
10. Other serious conditions that may limit patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2022-09-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 90 days post infusion
  Incidence of dose-limiting toxicities
The occurrence of AEs and SAEs during the study treatment | 0 to 28 days post infusion
  An adverse event is any undesirable experience associated with the use of a medical product in a patient

SECONDARY OUTCOMES:
Objective remission rate(ORR) | 1 year post infusion
  Imaging assessment of tumor remission
Progression free survival(PFS) | 2 year post infusion
  Progress Free Survival after administration
Overall survival (OS) | 2 years post infusion
  overall survival refers to the period from being included in the test group to death caused by any reason

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No